CLINICAL TRIAL: NCT00428844
Title: A Phase 2 Randomized Study Investigating the Safety, Efficacy and Pharmacokinetics of Daptomycin 6 mg/kg and 8 mg/kg Versus Comparator in the Treatment of Subjects Undergoing Surgical Standard of Care for Osteomyelitis Associated With an Infected Prosthetic Hip or Knee Joint Caused by Staphylococci
Brief Title: Study of Daptomycin in Subjects Undergoing Surgery for Osteomyelitis Associated With an Infected Prosthetic Caused by Staphylococci
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3009-016; DAP-OST-06-02 (Other: Cubist Study Number)
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Osteomyelitis
Keywords: Osteomyelitis; Prosthetic Hip; Prosthetic Knee; MRSA; Osteomyelitis Associated with an Infected Prosthetic Hip or Knee Joint; Staphylococci
MeSH Terms: conditions — Osteomyelitis | interventions — Daptomycin; Vancomycin; Teicoplanin; Nafcillin; Oxacillin; Floxacillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Daptomycin 6 mg/kg (Experimental): Daptomycin (6 mg/kg every 24 hours [q24h]) as a 30 minute intravenous (IV) infusion for 6 weeks (± one week).
  Interventions: Drug: daptomycin
- Daptomycin 8 mg/kg (Experimental): Daptomycin (8 mg/kg q24h) as a 30 minute IV infusion for 6 weeks (± one week).
  Interventions: Drug: daptomycin
- Comparator (Active Comparator): Vancomycin was administered at 1 gram every 12 hours (q12h) as a 60-minute infusion and teicoplanin was administered 6 mg/kg q24h as a 30-minute infusion also for 6 weeks (±1 week). Semi-synthetic penicillin (nafcillin, oxacillin, or flucloxacillin) was administered according to standard of care for 6 weeks (±1 week).
  Interventions: Drug: vancomycin; Drug: teicoplanin; Drug: nafcillin; Drug: oxacillin; Drug: flucloxacillin

INTERVENTIONS:
Drug: daptomycin — 6 mg/kg
  Other Names: Cubicin
  Arms: Daptomycin 6 mg/kg
Drug: daptomycin — 8 mg/kg
  Other Names: Cubicin
  Arms: Daptomycin 8 mg/kg
Drug: vancomycin — 1 gram
  Other Names: Vancocin
  Arms: Comparator
Drug: teicoplanin — 6 mg/kg; used only at UK sites
  Other Names: Targocid
  Arms: Comparator
Drug: nafcillin — 1-2 gram
  Other Names: Unipen
  Arms: Comparator
Drug: oxacillin — 1-2 gram
  Other Names: Bactocill
  Arms: Comparator
Drug: flucloxacillin — 1-2 mg
  Other Names: Fluclox
  Arms: Comparator

SUMMARY:
This is a research study designed to look at the efficacy and safety of daptomycin given at a dose of 6 mg/kg or 8 mg/kg in subjects being treated for prosthetic hip or knee infections caused by Staphylococci. These types of bacteria are among the most common types of bacteria causing infections of prosthetic joints.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between the ages of 18 and 80, inclusive
* Subject must have a diagnosis of prosthetic joint infection (PJI) in a hip or knee joint which has never previously been totally revised because of an infection and for which they are anticipated to undergo a two-stage replacement surgery
* Subject must have a positive microbiological identifier of staphylococci.
* If Subject is female of childbearing potential, must be willing to practice reliable birth control

Exclusion Criteria:

* Subject has permanent intravascular prosthetic material such as heart valves or pacemakers
* Subject has a creatinine clearance (CLCR) <30 mL/min as determined by the Cockcroft-Gault equation using actual body weight.
* Subject has significant hepatic dysfunction
* Subject has a fungal or mycobacterial PJI
* Subject is known to be HIV-infected with CD4 count ≤ 200 cells/ mm3
* Subject has an abnormal creatine phosphokinase (CPK) (elevated CPK level ≥ 2x ULN) at baseline as measured by central laboratory
* Subject is currently under treatment with chemotherapeutic agents excluding chronic maintenance therapy (e.g. tamoxifen to prevent relapse of primary breast cancer)
* Subject is pregnant, nursing, or lactating.
* Subject is receiving or is expected to receive chronic immunosuppressive therapy during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-06-26 (Actual); Primary Completion 2010-03-26 (Actual); Study Completion 2010-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alistair Wheeler, MD, Study Director — Cubist Pharmaceuticals, 65 Hayden Ave, Lexington, MA 02421, USA
Locations (26):
- United States (17):
  - UAMS College of Medicine, Little Rock, Arkansas
  - South Denver Infectious Disease Associates, PC, Englewood, Colorado
  - Kane and Davis Associates, Washington D.C., District of Columbia
  - Infectious Disease Association of Tampa Bay, Tampa, Florida
  - Idaho Falls Infectious Diseases, PLLC, Idaho Falls, Idaho
  - Rush St. Luke's Medical Center, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Sierra Infectious Disease, Reno, Nevada
  - Dartmouth-Hitchcock Medical center, Lebanon, New Hampshire
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health Systems, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Regional Infectious Diseases-Infusion Center, Lima, Ohio
  - Lehigh Valley Hospital Trauma and Critical Care Research, Allentown, Pennsylvania
  - Rothman Institute, Philadelphia, Pennsylvania
  - Gundersen Clinic, LTD, La Crosse, Wisconsin
- Russia (6):
  - Federal National Institution of Science "Russian Ilizarov Scientific Center" "Restorative Traumatology and Orthopedics" of Rosmedtechnology, Kurgan
  - National Healthcare Institution of Moscow "City Clinical Hospital #64", Moscow
  - Federal Healthcare Institute "Novosibirsk Scientific Research Institute of Traumatology and Orthopedy Rosmeditechnology", Novosibirsk
  - National Educational Institution of Higher Professional Education "Saint Petersburg State Medical Academy n.a. Mechnikov of Roszdrav", Saint Petersburg
  - Russian Research Institute of Traumatology and Orthopedy, Saint Petersburg
  - National Healthcare Institution "Samara Regional Clinical Hospital n.a. Kalinin", Samara
- United Kingdom (3):
  - Nuffield Orthopaedics Centre, Bone Infection Unit, Headington, Oxford, Oxfordshire
  - The Royal Infirmary of Edinburgh at Little France, Edinburgh, Scotland
  - Brownlee Centre - Gartnavel General Hospital, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Byren I, Rege S, Campanaro E, Yankelev S, Anastasiou D, Kuropatkin G, Evans R. Randomized controlled trial of the safety and efficacy of Daptomycin versus standard-of-care therapy for management of patients with osteomyelitis associated with prosthetic devices undergoing two-stage revision arthroplasty. Antimicrob Agents Chemother. 2012 Nov;56(11):5626-32. doi: 10.1128/AAC.00038-12. Epub 2012 Aug 20. PMID 22908174

RESULTS

PARTICIPANT FLOW:
Groups:
- Comparator: Vancomycin was administered at 1 gram (gm)every 12 hours (q12h) as a 60-minute infusion and teicoplanin was administered 6 mg/kg q24h as a 30-minute infusion also for 6 weeks (±1 week). Semi-synthetic penicillin (nafcillin, oxacillin, or flucloxacillin) was administered according to standard of care for 6 weeks (±1 week).
Period: Completed Study Drug Treatment
Arm/Group | Daptomycin 6 mg/kg | Daptomycin 8 mg/kg | Comparator
Started | 25 | 24 | 26
Received First Dose | 25 | 24 | 25
Completed | 23 | 18 | 19
Not Completed | 2 | 6 | 7
Not completed — Adverse Event | 2 | 4 | 4
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Randomized Not Treated | 0 | 0 | 1
Period: Completed Test of Cure (TOC) Visit
Arm/Group | Daptomycin 6 mg/kg | Daptomycin 8 mg/kg | Comparator
Started | 23 | 18 | 19
Completed | 20 | 16 | 17
Not Completed | 3 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Microbiologic failure | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Daptomycin 6 mg/kg: Daptomycin (6 mg/kg q24h) as a 30-minute IV infusion for 6 weeks (±1 week).
- Daptomycin 8 mg/kg: Daptomycin (8 mg/kg q24h) as a 30-minute IV infusion for 6 weeks (±1 week).
- Comparator: Vancomycin was administered at 1 gm q12h as a 60-minute infusion and teicoplanin was administered 6 mg/kg q24h as a 30-minute infusion also for 6 weeks (±1 week). Semi-synthetic penicillin (nafcillin, oxacillin, or flucloxacillin) was administered according to standard of care for 6 weeks (±1 week).
- Total: Total of all reporting groups
Arm/Group | Daptomycin 6 mg/kg | Daptomycin 8 mg/kg | Comparator | Total
Number analyzed (Participants) | 25 | 24 | 25 | 74
Age, Categorical [Count of Participants; unit: Participants] — Safety/Intent to Treat Population (1 patient included in the Overall Number of Baseline Participants was randomized to comparator but not treated)
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 10 | 14 | 15 | 39
    >=65 years | 15 | 10 | 10 | 35
Sex: Female, Male [Count of Participants; unit: Participants] — Safety/Intent to Treat Population (1 patient included in the Overall Number of Baseline Participants was randomized to comparator but not treated)
  Participants
    Female | 14 | 10 | 11 | 35
    Male | 11 | 14 | 14 | 39

OUTCOME MEASURES:

1. Primary Outcome: Any Creatine Phosphokinase (CPK) Elevation > 500 Units Per Liter (U/L)
Description: Number of subjects with CPK >500 U/L between Day 3 and 7 days following the last dose of study medication (Day 7P) as measured by the central laboratory.
Time Frame: From the 3rd day of therapy to 1 week post last dose (approximately week 7)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Daptomycin 6 mg/kg | Daptomycin 8 mg/kg | Comparator
Number analyzed (Participants) | 25 | 24 | 25
Participants | 4 | 5 | 2

2. Secondary Outcome: Safety - Notable Laboratory Abnormalities
Description: Summary of Notable Laboratory Abnormalities - description of the proportion of subjects within each treatment group that had clinical laboratory values outside the reference range.
Time Frame: From the 1st day of therapy to maximum of 23 weeks post last dose (up to maximum of week 30)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Daptomycin 6 mg/kg | Daptomycin 8 mg/kg | Comparator
Number analyzed (Participants) | 25 | 24 | 25
Participants
  Hematocrit (<30%, >60%) | 12 | 10 | 15
  Hemoglobin (<9,>19 g/dL) | 10 | 10 | 12
  Red Blood Cell (Female <2.5,>6.0; Male <3.0, >6.5) | 2 | 4 | 3
  White Blood Cell (<2, >20 x 10^9/L) | 1 | 0 | 0
  Platelets (<40, >450 x 10^9/L) | 13 | 13 | 10
  Albumin (<3, >6 g/dL) | 7 | 4 | 4
  Alkaline Phosphatase (>1350 U/L) | 0 | 0 | 0
  Alanine aminotransferase (>235 U/L) | 0 | 0 | 0
  Aspartate aminotransferase (>185 U/L) | 1 | 0 | 0
  Total bilirubin (>2.2 mg/dL) | 0 | 0 | 0
  Blood Urea Nitrogen (>50 mg/dL) | 2 | 0 | 1
  Creatinine (Female >2.0; Male>2.8 mg/dL) | 1 | 0 | 2

3. Secondary Outcome: Overall Clinical Outcome
Description: The sponsor determined overall clinical outcome based on blinded review of clinical, microbiological, and radiological response of the subject including, but not limited to, clinical signs and symptoms of PJI, microbiological assessments, radiographic findings, and surgical procedures performed. Subjects were a success if both clinical and microbiological responses were success. A subject who failed to respond clinically or microbiologically was a failure. If microbiological response was non-evaluable and/or clinical evaluation at TOC was not performed, the subject was non-evaluable.
Time Frame: Approximately 6 weeks post last dose (approximately week 12)
Population: Modified Intent-to-Treat Population. Six treated patients in the ITT population were not included in the mITT population, as they did not have confirmed baseline staphylococcal infection.
Measure: Number; unit: Participants
Arm/Group | Daptomycin 6 mg/kg | Daptomycin 8 mg/kg | Comparator
Number analyzed (Participants) | 24 | 23 | 21
Participants
  Success | 13 | 13 | 8
  Failure | 10 | 8 | 11
  Nonevaluable | 1 | 2 | 2

4. Secondary Outcome: Microbiological Response
Description: Sponsor's assessment of subject-level microbiological response at the test-of-cure visit for the modified Intent-to-Treat (mITT) population.
Time Frame: Approximately 6 weeks post last dose (approximately week 12)
Population: Modified Intent to Treat Population. Six treated patients in the ITT population were not included in the mITT population, as they did not have confirmed baseline staphylococcal infection.
Measure: Number; unit: Participants
Arm/Group | Daptomycin 6 mg/kg | Daptomycin 8 mg/kg | Comparator
Number analyzed (Participants) | 24 | 23 | 21
Participants
  Success | 12 | 12 | 8
  Failure | 8 | 3 | 6
  Non-evaluable | 4 | 8 | 7

5. Secondary Outcome: Pharmacokinetic Parameter: Maximum Plasma Concentration (Cmax)
Description: The pharmacokinetic (PK) parameters of daptomycin at steady state for the 6 mg/kg and 8 mg/kg dose groups. On treatment day 4, PK samples for daptomycin levels were to be obtained prior to start of daptomycin infusion (0 hr) and at 0.5 hr (end of infusion), 1-1.5 hr, 3-5 hr, 8-12 hr, and 24 hr after the start of daptomycin infusion.
Time Frame: Day 4 (steady state)
Population: Pharmacokinetic evaluable population. Pharmacokinetics not analyzed for the comparator group.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Daptomycin 6 mg/kg | Daptomycin 8 mg/kg
Number analyzed (Participants) | 22 | 20
µg/mL | 59.1 [22.5 to 156] | 92.3 [56.1 to 172]

6. Secondary Outcome: Pharmacokinetic Parameter: Area Under the Concentration-time Curve During a Dosing Interval at Steady State (AUCss)
Description: as for outcome 5
Time Frame: Day 4 (steady state)
Population: Pharmacokinetic evaluable population. Pharmacokinetics not analyzed for the comparator group.
Measure: Median (Full Range); unit: µg•hr/mL
Arm/Group | Daptomycin 6 mg/kg | Daptomycin 8 mg/kg
Number analyzed (Participants) | 22 | 20
µg•hr/mL | 499 [166 to 1205] | 821 [292 to 1606]

ADVERSE EVENTS:
Time Frame: From the 1st day of therapy to maximum of 23 weeks post last dose (up to maximum of week 30)
Description: Subjects who prematurely discontinue study drug will undergo follow-up safety evaluations within 30 days (±5 days) of administration of the last dose of study drug.
Arm/Group | Daptomycin 6 mg/kg | Daptomycin 8 mg/kg | Comparator
Serious Adverse Events (participants affected / at risk) | 8/25 | 4/24 | 8/25
Other Adverse Events (participants affected / at risk) | 23/25 | 18/24 | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin 6 mg/kg (N=25) | Daptomycin 8 mg/kg (N=24) | Comparator (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Wound necrosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin 6 mg/kg (N=25) | Daptomycin 8 mg/kg (N=24) | Comparator (N=25)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3) | 4 (7)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (5)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Catheter related complication (General disorders) | 1 (1) | 2 (3) | 2 (9)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (3)
Oedema peripheral (General disorders) | 2 (5) | 2 (4) | 4 (7)
Pyrexia (General disorders) | 4 (5) | 2 (2) | 4 (7)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Bacteriuria (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 2 (2) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 3 (5) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication is initiated by Cubist. If first publication not published within 1 year of study conclusion or termination, Investigator has right to publish and disclose the Data. Prior to any submission for publication, presentation, or communication of results or information arising from the Study, Investigator shall provide Cubist at least 90 days for review and comment upon the manuscript or other material for such publication or presentation.